CLINICAL TRIAL: NCT01761110
Title: Development of a Community-based Buprenorphine Treatment Intervention
Brief Title: Pilot Test of a Community-based Buprenorphine Treatment Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); City University of New York (Other); Washington Heights Corner Project (Unknown)
Responsible Party: Principal Investigator, Chinazo Cunningham, Professor, Albert Einstein College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-381; R34DA031066 (NIH)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Opioid Dependence; Injection Drug Use
Keywords: Opioid dependence; Injection drug use; Buprenorphine; Opioid agonist treatment; Access to care; HIV risk behaviors; Opioids
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Participants will be enrolled prior to the implementation of the community-based buprenorphine treatment (CBBT) intervention.
- Post-intervention (Experimental): Participants will be enrolled after implementing the community-based buprenorphine treatment (CBBT) intervention
  Interventions: Behavioral: Community-based buprenorphine treatment (CBBT) intervention

INTERVENTIONS:
Behavioral: Community-based buprenorphine treatment (CBBT) intervention — Community-based buprenorphine treatment (CBBT) intervention consists of three components which are delivered to staff of syringe exchange programs, including: 1) providing buprenorphine education, 2) facilitating access to buprenorphine treatment, and 3) providing support to individuals who initiate buprenorphine treatment.
  Arms: Post-intervention

SUMMARY:
The main goal of this study is to pilot test the community-based buprenorphine treatment (CBBT) intervention, examining buprenorphine treatment initiation, opioid use, and HIV risk behaviors. Two groups of participants will be followed for 60 days, with 3 research visits. One group will be enrolled prior to the CBBT intervention (pre-intervention), and one group after the CBBT intervention (post-intervention). Data sources will include questionnaires, urine toxicology tests, and medical record data. Investigators hypothesize that compared to the participants in the pre-intervention group, participants in the post-intervention group will be more likely to initiate buprenorphine treatment, reduce opioid use, and reduce high-risk HIV risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* English or Spanish fluency
* ever injected drugs
* not receiving buprenorphine treatment (no prescribed buprenorphine in the previous 6 months)
* clients of our collaborating community-based organization
* interested in buprenorphine treatment

Exclusion Criteria:

* pregnant
* taking more than 60mg of methadone daily in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
initiation of buprenorphine treatment | 60 days
  Medical record information will be extracted to determine initiation of buprenorphine treatment, which will be defined as a visit with a medical provider in which buprenorphine is prescribed.

SECONDARY OUTCOMES:
opioid use | 60 days
  Opioid use will be determined via self-report using the Addiction Severity Index and via urine specimens (e.g., urine toxicology testing).

OTHER OUTCOMES:
HIV risk behaviors | 60 days
  Drug- and sex-related HIV risk behaviors will be assessed using a standardized risk assessment tool used in NIDA's Clinical Trials Network.

CONTACTS AND LOCATIONS:
Overall Officials: Chinazo Cunningham, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Washington Heights Corner Project, New York, New York, United States